CLINICAL TRIAL: NCT06638203
Title: The Effect of "NurseLead in Progress" Game on the Development of Transformational Leadership Behaviors of Nursing Students: A Randomized Controlled Study
Brief Title: The Effect of a Game on the Development of Leadership Behaviors of Nursing Students
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canberk Akdeniz (Other)
Responsible Party: Sponsor-Investigator, Canberk Akdeniz, Principal Investigator. PhD Candidate at Hacettepe University Institute of Health Sciences, Türkiye, enrolled in the Nursing Fundamentals and Management Integrated PhD Program., Hacettepe University
Organization: Hacettepe University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: E-66777842-300-00003535955
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Leadership
Keywords: Computer Games; Leadership; Nursing Students; Role Playing; Randomized Controlled Trial

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Expert A will assess the students' eligibility based on predetermined inclusion and exclusion criteria. From those who qualify, Expert B will use specialized software to randomly select 50 participants through systematic random sampling. An independent Expert C will then randomly assign these 50 students to either the control or intervention groups using block randomization. Expert D will administer the pre- and post-tests, which will then be sent to statisticians for analysis. After the statistical results are received and reported, the researchers will know which students were in the control or intervention group. The intervention group will participate in the game first, while the control group will be placed on a waitlist and will play the game after the statistical analysis is completed. Although the control group will also have the opportunity to develop their leadership skills through the game, their performance will not be evaluated post-play.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants who will complete the leadership course and then engage in the leadership game
  Interventions: Other: The 2-hour Exemplary Leadership Course (ELC); Other: The NurseLead in Progress Game
- Control Group (Active Comparator): Participants who will complete the leadership course only.
  Interventions: Other: The 2-hour Exemplary Leadership Course (ELC)

INTERVENTIONS:
Other: The 2-hour Exemplary Leadership Course (ELC) — This two-hour course, based on the Five Exemplary Leadership Model, aims to refresh participants' theoretical understanding of leadership while providing insights into effective leader-follower interactions through practical scenarios. The session will begin with an exploration of the nature of leadership, including its philosophical and historical context. The significance of leadership in nursing will be emphasized, highlighting its impact on education, clinical practice, and the profession overall. Participants will examine the key roles of nurse leaders, focusing on modeling the way, inspiring a shared vision, challenging the process, enabling others to act, and encouraging the heart. Content Outline:
  1. The Nature and Definition of Leadership (5 minutes)
  2. Leadership and Its Importance in Nursing (15 minutes)
  3. Transformational Leadership and Its Components (40 minutes)
  4. Positive Leader-Follower Interactions (15 minutes)
  5. Case Study Discussions (45 minutes)
Other: The NurseLead in Progress Game — Developed collaboratively by the author and a company, this unpublished game focuses on role-playing leader-follower interactions to navigate scenarios effectively. Designed for five students per session, the game consists of five sections, lasting approximately one hour, with each section corresponding to one of the Five Practices of Exemplary Leadership. In each section, one student takes on the role of leader while the other four act as followers. The main objective is to guide a newly appointed charge nurse in making sound decisions when facing challenges to achieve key goals. Following the game, a debriefing session will allow participants to analyze responses with experts. Performance will not be formally evaluated, as the game serves as a learning experience, enabling students to lead and engage as followers. This activity aims to activate the experiential learning phase of Kolb's Learning Model.
  Arms: Intervention Group

SUMMARY:
The aim of this randomized controlled trial is to examine the effect of a leadership role-playing computer game on nursing students' leadership practices. The main questions it aims to answer are:

RQ1: Will participants in the intervention group perform better on the Five Practices of Exemplary Leadership Achievement Test (5PELAT) after the game?

* RQ1a: Is the average score of the intervention group on the Five Practices of Exemplary Leadership Achievement Test significantly higher than the average score of the control group after the game?
* RQ1b: Is the difference between pre-test and post-test scores on the Five Practices of Exemplary Leadership Achievement Test significantly greater in the intervention group compared to the control group?

RQ2: Will participants in the intervention group report higher self-assessments of their own leadership practices after the game compared to the control group?

* RQ2a: Is the average score of the intervention group on the Student Leadership Practices Inventory (SLPI) significantly higher than the average score of the control group after the game?
* RQ2b: Is the difference between pre-test and post-test scores on the Student Leadership Practices Inventory significantly greater in the intervention group compared to the control group?

Researchers will compare the leadership course & game playing intervention to only getting the leadership course to see if the combined version works better in developing nursing students' transformational leadership. Participants will:

* Take the leadership course and play the leadership game or only take the course.
* Complete Five Practices of Exemplary Leadership Achievement Test (5PELAT) and the Student Leadership Practices Inventory (SLPI) before and after the intervention.

DETAILED DESCRIPTION:
Study Design The study is planned as a parallel group randomized controlled study to determine the effect of the "NurseLead in Progress" computer game on subjective and objective leadership measurement. At the end of the study, it is aimed to evaluate the effect of getting the leadership course only to combining it to a role-playing involved gameplay. The experiment will not measure the effectiveness of the game intervention, but its efficacy under ideal conditions. In this context, an explanatory design will be used. Since the number of participants was previously calculated in the light of reference articles, a fixed design will be used in terms of the number of participants. CONSORT 2024 will be used for reporting the research.

Settings and Participants The course and the game intervention will take place in the office of a nursing union, a central location based in Ankara/Türkiye. The population is the nursing students in Ankara/Türkiye as well. In Ankara, there are 4 public and 6 private universities that gives 4 years BSN education and total number of nursing students is nearly 5000. Based on the lowest effect size in the reference articles (Foli et al, 2014; Marath & Ramachandra, 2015) it was calculated that there should be 18 students in the groups with a ratio of n intervention/ n control=1 to provide 80% power, 0.99 effect size (Cohen's) and 2.5% Type I error (One-way hypothesis) in order to compare two independent group averages. In order to reach the largest sample size to test all hypotheses, it was planned to include 25 students each in the intervention and control groups with an estimated 25% dropout rate in the groups, considering the long-term data collection phase and the variability in motivation to participate in extracurricular activities. The inclusion and exclusion criteria is mentioned elsewhere. The nursing students meet the inclusion criteria will be informed about the purpose, content and method of the study and the sample group (experimental and control) will be formed by obtaining written permission from those who voluntarily agree to participate in the study. Determination of the experimental and control groups will be provided by https://www.randomizer.org/ website.

Instruments Author prepared Introductory Information Form will be used to investigate baseline comparisons. Author-prepared Five Practices of Exemplary Leadership Achievement Test (5PELAT) will be used to collect objective data on the leadership development. In addition, Student Leadership Practices Inventory (SLPI), by Kouzes and Posner will be used to collect nursing students' perspective on their leadership development.

The Introductory Information form consists of two parts. The first part includes 10 questions about students' individual and academic characteristics and the second part includes 10 questions about their participation in professional activities.

Five Practices of Exemplary Leadership Achievement Test consists of 10 questions, each with five options, on a sample scenario, analyzed according to the Five Practices of Exemplary Leadership model. It will be administered to all participants in the pre-test and post-test in order to provide an objective assessment of the change in leadership behaviors. The questions have been prepared together with experts and finalized with the opinions of a widely participated expert panel.

The Student Leadership Practices Inventory, developed by Kouzes and Posner for undergraduate students to assess their own leadership practices, has 5 sub-dimensions. The sub-dimensions of the inventory, which consists of 30 questions in total, are modeling the way, inspiring a shared vision, challenging the process, enabling others to act and, and encouraging the heart. The 5-point Likert scale has no reverse items. There are 6 questions for each sub-dimension. The scores that can be obtained from each sub-dimension are between 6-30. The total score that can be obtained from the scale is between 30-150. The higher the score obtained from the scale, the more positive the students' attitude towards their own leadership practices. It is planned to be applied as a pre and posttest to measure the participants' evaluations of their leadership behaviors. The inventory will be applied in Turkish format and the related adaptation study was carried out by the authors and presented as an oral presentation at the 8th International 19th National Nursing Congress at Hacettepe University Sıhhiye Cultural Center on September 25-28, 2024. Cronbach's alpha coefficient for the self-assessment version to be used in the experiment was .959. The CVR values were above 0.9 and each CVI for the sub-dimensions was above 0.97. In confirmatory factor analysis, all factor loads were above 0.30.

Data Collection

Pre-Randomization Before randomization, we will invite all eligible students to participate in the study by signing a voluntary consent form. An independent expert (A), not affiliated with the research team, will assess the students' eligibility based on inclusion and exclusion criteria. From those who meet the criteria, another independent expert (B) will use appropriate software to randomly select 50 participants through systematic random selection.

Randomization and Blinding An independent expert (C) will randomly allocate the 50 selected students into control and intervention groups using block randomization. Blinding process is detailed in elsewhere.

Consent Collection and Leadership Course Implementation We will provide all participating students (n=50) with Voluntary Consent Forms and ask them to return the signed forms. Following this, we will conduct a 2-hour Leadership Training Program. The program aims to refresh participants' theoretical knowledge of leadership, offer insights into key elements for effective leader-follower interactions, and ensure that all participants have a similar level of theoretical understanding and practical potential before the intervention. Additionally, the program will include case study discussions based on the Exemplary Leadership Framework.

Administration of Introductory Information Form and Pre-Test All students who complete the training program will fill out the introductory form, which is designed to identify any initial differences. At the same time, each participant will take the Five Practices of Exemplary Leadership Achievement Test and the Student Leadership Practices Inventory.

Game Implementation After completing the course, participants in the intervention group will engage in the game. Designed for five students per session, the game consists of five sections and lasts approximately one hour. Each section aligns with one of the Five Practices of Exemplary Leadership. In each section, one student will assume the role of the leader, while the other four act as followers. The game's main objective is to guide a newly appointed charge nurse in making the right decisions when faced with challenges, ultimately achieving the final goals. After the game, a debriefing session will be held, where responses will be analyzed with experts and students. Performance in the game will not be formally measured, as it is purely a learning experience designed to provide opportunities for students to lead and effectively share as followers. The game is intended to activate the experiential learning phase of Kolb's Learning Model.

Post-Test Two weeks after the intervention group completes the game and feedback sessions, the post-test will be administered. Both the intervention and control groups will take the achievement test and the Student Leadership Practices Inventory. The achievement test in this phase will be identical in scenario and questions to the first test.

Data Analysis The data will be analyzed using the SPSS 25.0 package program. The descriptive characteristics of the participants will be analyzed using means and standard deviations for continuous variables and frequencies and percentages for categorical variables. Differences in characteristics between the intervention and control groups will be analyzed using independent t-tests or chi-square tests. In addition, the initial comparability of the groups, i.e. the success of random assignment, will be statistically tested. Paired t-tests will be used to analyze within-group outcome differences between the pretest and posttest. For one-way hypothesis tests, all results with p<.025 will be considered statistically significant. ITT and PP analyses will be used to analyze the data of the participants who were separated from the control and intervention groups within the sample. If the characteristics of the data are appropriate, analyses such as cox regression, Manova, multivariate regression, two-way analysis of variance in repeated measures will also be performed to analyze whether the outcome is caused by the intervention (causality).

Ethical Considerations Ethical approval was obtained from Hacettepe University's Social Sciences and Humanities Researches Ethics Board. Additionally, permission was secured from Kouzes and Posner for the adaptation of the leadership inventory, and approval for its use was granted by Wiley. Institutional permissions were obtained from the relevant union for the office where the intervention will take place. Participation in the game development and gameplay will be free of charge for the participants. Furthermore, their travel expenses to the office where the trial will be conducted will be covered by Researcher #1. Participants within each group will be selected from different universities, ensuring that no group consists of students from the same institution.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between 18 and 25 years old.
* Informed consent must be obtained from the participant.
* Participants must have no visual and/or hearing impairments.
* Participants must be students in a four-year nursing bachelor's program.
* Participants must be in the 3rd or 4th year of their bachelor's program.
* Participants must have completed a leadership course during their bachelor's education.

Exclusion Criteria:

* Individuals who are younger than 18 or older than 25 years old.
* Individuals with visual and/or hearing impairments.
* Individuals who are currently receiving or have received training related to leadership outside of their program.
* Individuals holding a diploma in a field other than nursing.
* Individuals currently studying in a field other than nursing.
* Individuals who have suspended their bachelor's education.
* Individuals who are in the preparatory year, 1st, or 2nd year of the bachelor's program.
* Individuals who have not taken any leadership-related courses during their bachelor's education.
* Individuals with a conflict of interest due to close relationships with the researchers.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Transformational Leadership Development (Objective) | Before the interventions, in both groups (baseline) 2 weeks after the interventions, in both groups. (1st measurement) 4 weeks after the interventions, in both groups. (2nd measurement) In total, time frame is 6 weeks.
  Five Practices of Exemplary Leadership Achievement Test (5PELAT)
  The 5PELAT is a test developed by the authors, comprising 10 questions, each featuring 5 response options based on various sample scenarios. These scenarios are analyzed in alignment with the Five Practices of Exemplary Leadership model. Each question and its corresponding answers have been crafted in collaboration with subject matter experts and refined through feedback from an expert panel, ensuring their relevance and effectiveness in evaluating leadership. This development process aims to provide reliable insights into participants' understanding and application of exemplary leadership practices.

SECONDARY OUTCOMES:
Transformational Leadership Development (Perspective) | Before the interventions, in both groups (baseline) 2 weeks after the interventions, in both groups. (1st measurement) 4 weeks after the interventions, in both groups. (2nd measurement) In total, time frame is 6 weeks.
  The Student Leadership Practices Inventory (SLPI-Self)
  The SLPI developed by Kouzes and Posner for students to assess their own leadership practices, has 30 items (no reverse coding) and 5 sub-dimensions. There are 6 questions for each sub-dimension. The scores that can be obtained from each sub-dimension are between 6-30. The total score that can be obtained from the scale is between 30-150. The higher the score obtained from the scale, the more positive the students' attitude towards their own leadership practices.

CONTACTS AND LOCATIONS:
Overall Officials: Canberk Akdeniz, Principal Investigator — HEP-SEN Union (Senior Advisor); Sergül Duygulu, Prof., Study Director — Hacettepe University Nursing Faculty
Locations (1):
- HEP-SEN Union - Ankara Prof. Dr. Perihan Velioglu Branch, Ankara, Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
We intend to upload the raw, de-identified data to Mendeley Data. The publication of the dataset will be contingent upon the manuscript's publication, following the completion of all necessary processes.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Beginning 1 year after publication with no end date
Access Criteria: Individual participant data (IPD) will be made available upon request to researchers-excluding those affiliated with or funded by a company-who wish to conduct a systematic review, meta-analysis, or sample size calculations. Only the inventory scores (including score values but not item details-due to Wiley requirements) will be shared. Researchers seeking access to the IPD must contact both authors, and both must provide consent for data sharing.

REFERENCES:
- [Background] Tunn R, Boutron I, Chan AW, Collins GS, Hrobjartsson A, Moher D, Schulz KF, de Beyer JA, Hansen Nejstgaard C, Ostengaard L, Hopewell S. Methods used to develop the SPIRIT 2024 and CONSORT 2024 Statements. J Clin Epidemiol. 2024 May;169:111309. doi: 10.1016/j.jclinepi.2024.111309. Epub 2024 Feb 29. PMID 38428538
- [Background] Marath, U., Ramachandra, (2015). Impact of Leadership Development Package on Leadership Competencies of Undergraduate Nursing Students. Asian J. Nur. Edu. and Research 5(2): April-June 2015; Page221-228. doi: 10.5958/2349-2996.2015.00044.0
- [Background] Kuruca Ozdemir E, Dinc L. Game-based learning in undergraduate nursing education: A systematic review of mixed-method studies. Nurse Educ Pract. 2022 Jul;62:103375. doi: 10.1016/j.nepr.2022.103375. Epub 2022 Jun 13. PMID 35749962
- [Background] Kouzes, James M., Barry Z. Posner. (2017). The Leadership Challenge 6th ed. Hoboken, NJ: Wiley.
- [Background] Kouzes, James M., Barry Z. Posner. (2013). The Student Leadership Challenge: Facilitation and Activity Guide. San Francisco: Jossey-Bass.
- [Background] Kolb, D.A. (1984) Experiential Learning: Experience as the Source of Learning and Development. Englewood Cliffs, N.J.: Prentice-Hall
- [Background] Foli KJ, Braswell M, Kirkpatrick J, Lim E. Development of leadership behaviors in undergraduate nursing students: a service-learning approach. Nurs Educ Perspect. 2014 Mar-Apr;35(2):76-82. doi: 10.5480/11-578.1. PMID 24783721
- [Background] Denney, Logan R., "Student Leadership Development: A Focus on Experiential Leadership Orientation Within Higher Education" (2013). Master of Arts in Higher Education (MAHE) Theses. 94. https://pillars.taylor.edu/mahe/94
- [Background] Petit dit Dariel OJ, Raby T, Ravaut F, Rothan-Tondeur M. Developing the Serious Games potential in nursing education. Nurse Educ Today. 2013 Dec;33(12):1569-75. doi: 10.1016/j.nedt.2012.12.014. Epub 2013 Jan 16. PMID 23332500
- [Background] Curtis EA, de Vries J, Sheerin FK. Developing leadership in nursing: exploring core factors. Br J Nurs. 2011 Mar 10-23;20(5):306-9. doi: 10.12968/bjon.2011.20.5.306. PMID 21471879
- [Background] Boctor L. Active-learning strategies: the use of a game to reinforce learning in nursing education. A case study. Nurse Educ Pract. 2013 Mar;13(2):96-100. doi: 10.1016/j.nepr.2012.07.010. Epub 2012 Aug 19. PMID 22910398
- [Background] Blakely G, Skirton H, Cooper S, Allum P, Nelmes P. Educational gaming in the health sciences: systematic review. J Adv Nurs. 2009 Feb;65(2):259-69. doi: 10.1111/j.1365-2648.2008.04843.x. Epub 2008 Nov 14. PMID 19032512
- [Background] Akdeniz C, Duygulu S. Systematic Review on Characteristics and Effects of Leadership Development Interventions for Nursing Students. Nurse Educ. 2024 May-Jun 01;49(3):E147-E152. doi: 10.1097/NNE.0000000000001540. Epub 2023 Nov 16. PMID 37994497